CLINICAL TRIAL: NCT06735157
Title: Repetitive Transcranial Magnetic Stimulation Paired with Augmented Reality to Alter Concussion Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Greenbank Concussion Clinic (Unknown)
Responsible Party: Principal Investigator, Aimee Nelson, Aimee J. Nelson, PhD, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17699
Record Dates: First submitted 2024-12-10; First posted 2024-12-16 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Mild Traumatic Brain Injury, Concussion; Chronic Dizziness; Vestibular Problem
Keywords: Concussion; Dizziness; Transcranial magnetic stimulation; augmented reality; repetitive transcranial magnetic stimulation; mild traumatic brain injury; intermittent theta burst stimulation; accelerated iTBS; balance training; vestibular rehabilitation therapy
MeSH Terms: conditions — Brain Concussion; Vestibular Diseases; Dizziness | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be split into two groups, one that will receive real rTMS and one that will receive sham rTMS.
Who Masked: Participant
Masking Description: Participants will be blinded to their intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham rTMS (Sham Comparator)
  Interventions: Behavioral: Augmented reality vestibular rehabilitation therapy; Device: SHAM repetitive transcranial magnetic stimulation
- Real rTMS (Active Comparator)
  Interventions: Device: Repetitive transcranial magnetic stimulation; Behavioral: Augmented reality vestibular rehabilitation therapy

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Repetitive transcranial magnetic stimulation (intermittent theta burst stimulation) will be delivered using a Magstim Rapid 2 stimulator (Magstim, Whitland, UK) guided using neuronavigation (Brainsight, Rogue Research, Montreal, QC, Canada) to target primary motor cortex. Participants will receive 14 days of stimulation over a 3-week period. Stimulation will use a protocol called accelerated iTBS (Duprat et al., 2016) whereby iTBS will be delivered three times during the same study session. Each iTBS session will deliver 600 pulses in 50 Hz bursts of 3 pulses for a total of 1800 pulses delivered each day. iTBS sessions will each be separated by 15 minutes (Duprat et al., 2016; Wu et al., 2013). Stimulation will be delivered at 70% of the participant's resting motor threshold. Immediately following each 600-pulse period of iTBS, individuals will participate in 5 to 10 minutes of AR vestibular rehabilitation therapy.
  Other Names: Intermittent theta burst stimulation
  Arms: Real rTMS
Behavioral: Augmented reality vestibular rehabilitation therapy — Participants will complete the vestibular training through Nreal Air AR Glasses (Nreal, China). The vestibular training task was custom-made in Unity V2021.3.14fI software using C+ script language. Participants will be standing upright for the AR training, with a safety bar positioned directly in front of them should they need to hold onto something. A large cross-shaped target will be positioned approximately 3 feet in front of the participant's head with its vertical center aligned with the participant's midline. This will act as a visual starting point. The training is adapted from clinical vestibular rehabilitation training methods used in PCD. The vestibular training task consists of locating and tracking a series of moving 3-dimensional balls presented at random within the participant's field of view.
  Other Names: Vestibular rehabilitation therapy; Balance training; Vestibular training; Augmented reality
Device: SHAM repetitive transcranial magnetic stimulation — Sham repetitive transcranial magnetic stimulation will be delivered using a Magstim Rapid 2 sham stimulator (Magstim, Whitland, UK) guided using neuronavigation (Brainsight, Rogue Research, Montreal, QC, Canada) to target primary motor cortex. Participants will receive 14 days of sham stimulation over a 3-week period. Stimulation will use a protocol called accelerated iTBS (Duprat et al., 2016) whereby sham iTBS will be delivered three times during the same study session. Each sham iTBS session will sound and feel identical to real iTBS delivery, but will not deliver a stimulating current. Sham iTBS sessions will each be separated by 15 minutes (Duprat et al., 2016; Wu et al., 2013). Sham stimulation will be delivered at 70% of the participant's resting motor threshold. Immediately following each 600-pulse period of sham iTBS, individuals will participate in 5 to 10 minutes of AR vestibular rehabilitation therapy.
  Other Names: Sham intermittent theta burst stimulation
  Arms: Sham rTMS

SUMMARY:
This study aims to determine whether the delivery of brain stimulation paired with a balance training task can improve symptoms of dizziness for individuals experiencing these symptoms due to concussion. The main questions it aims to answer are:

* Does repetitive transcranial magnetic stimulation (rTMS) paired with balance training improve the symptoms of dizziness in individuals with persistent dizziness due to concussion?
* Is the proposed rTMS and balance training protocol feasible in this population?

Researchers will compare results from a sham rTMS group with those from a real rTMS group to see if any observed changes are from the placebo effect rather than the expected effects of real rTMS.

Participants will receive pulses of rTMS to the area of the brain responsible for control of movement and then be asked to interact with digital objects using augmented reality glasses for 14 days over 3 weeks.

DETAILED DESCRIPTION:
The incidence of traumatic brain injury (TBI) is increasing in Canada, and it is expected to be one of the most common neurological conditions affecting Canadians by 2031. Up to 90% of TBIs are classified as mild (m)TBI, also known as concussion. A federal concussion report from 2019 indicated an annual prevalence of 200,000 mTBIs in Canada. Symptoms of mTBI, termed post-concussion symptoms (PCS), include dizziness, headache, alterations in mood, and cognitive impairment. PCS generally resolves on its own. However, some patients experience persistent PCS lasting beyond 3 months after the initial head injury.

Dizziness is the second most common symptom of mTBI after headache. It is estimated that up to 81% of mTBI patients will present with dizziness upon initial clinical examination, which may continue to persist beyond 1-year following the initial trauma in 25% of patients. Post-concussion dizziness (PCD) can present as postural instability, ongoing vertigo, balance impairments, nausea, and intolerance to head motion. These symptoms can drastically reduce quality of life and impact the ability to drive, work, and perform daily activities.

PCD is typically associated with vestibular impairment. Further, many patients complaining of dizziness following mTBI demonstrate physiologic abnormalities with the auditory and vestibular systems. Consequently, the most preferable treatment for PCD is a form of balance training called vestibular rehabilitation therapy (VRT). VRT consists of a set of exercises which promote adaptation, substitution, and habituation of the vestibular system. Adaptation, mediated by neuroplasticity, is the gradual remodelling of the nervous system as it "adapts" to the signals from the damaged vestibular system. Substitution is the process of learning strategies to compensate for poor vestibular function. Habituation is the gradual desensitization to certain movements through repeated exposure to those movements. These exercises are often individually prescribed based on personal areas of disability. Specific exercise types include gaze stability, habituation, substitution, and balance exercises. These target deficits in the vestibulo-ocular reflex (VOR), improve impaired motion sensitivity, facilitate central reprogramming, and improve balance. Traditional VRT, such as a balance task, is monotonous and often requires trained professionals to administer. VRT, in the form of interactive games, however, is engaging and has been shown to affect balance, dizziness, and mobility positively. A form of sensorimotor training consisting of an interactive game presented through augmented reality (AR) has not yet been explored. It may serve to reduce PCD by similar mechanisms as the aforementioned VRTs.

AR is typically presented through opaque glasses, which overlay virtual objects onto the user's environment. Users can then interact with both the virtual and physical environments simultaneously. Our AR intervention involves a game that promotes goal-directed movements of the head to accomplish tasks in various head orientations and postural positions. Through repeated exposure, this game aims to facilitate adaptation, substitution, and habituation of the vestibular system to reduce PCD.

A non-invasive neuromodulation technique called repetitive transcranial magnetic stimulation (rTMS) may improve AR vestibular training. One form of rTMS delivery called intermittent theta burst stimulation (iTBS) promotes synaptic plasticity by inducing long term potentiation (LTP)-like changes in neuronal excitability. Literature suggests that iTBS delivered to the primary motor cortex (M1) may improve learning in conjunction with motor training. rTMS may also improve dizziness. Ten sessions of rTMS reduce dizziness symptom severity and frequency by more than 50% in patients suffering from severe PCD. iTBS delivered to M1 improves balance in post-stroke patients. Systemic inflammation is an important physiological response to mTBI that may contribute to dizziness. Several studies have observed the anti-inflammatory effects of rTMS in clinical populations such as stroke and depression. Zhao et al. found that 20 sessions of rTMS on patients with refractory depression reduced elevated levels of TNF-⍺ and IL-1β to that of healthy controls. Levels of BDNF, which is important for brain growth, increased to that of healthy controls following the intervention. This effect on TNF-⍺, IL-1β, and BDNF was not observed in the clinical control group who did not receive rTMS. Cha et al. reported a similar reduction in inflammatory cytokines TNF-⍺, IL-1β, and IL-6 after 10 sessions of rTMS in post-stroke patients. Velioglu et al. found that 10 sessions of rTMS increased BDNF in patients with Alzheimer's disease. These effects also provide evidence towards a possible mechanism behind the effect of rTMS on other persistent PCS.

Patients with severe persistent PCD often require medical or surgical intervention. There is a clear need for non-invasive treatment options for these individuals. The primary objective of this study is to determine if the proposed technique is feasible and can be used to alter concussion symptoms in patients with PCD in a larger study. This study will also explore the effects of iTBS in combination with AR vestibular training on dizziness disability and postural stability in patients with PCD. Additionally, this research aims to determine if rTMS can modulate inflammation in persistent PCS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-65 years
* Diagnosis of mTBI according to the American Congress of Rehabilitation Medicine Diagnostic Criteria (Silverberg et al., 2023). All participants have diagnosis confirmed with Dr. Rathbone before enrollment.
* Persistent dizziness beyond 3-months following the initial head injury.
* Comprehension of spoken and written English language or have a language interpreter present for all study visits.

Exclusion Criteria:

* History of chronic dizziness unrelated to concussive events.
* Contraindications to TMS: presence of pacemaker, metal/electrical/magnetic implants not including titanium, known history of untreated or uncontrolled psychological disorders, pregnancy, history of seizure or diagnoses of epilepsy, taking medications that increase the risk of seizure.
* Inability to continue current medical therapies for the duration of the study.
* If imaging was done at the time of injury, individuals with a positive CT head will be excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory (DHI) | At baseline (before the first intervention session) and post-intervention (following the final intervention session)
  The DHI is a well-validated 25-item questionnaire which will be used to assess functional, physical, and emotional domains of disability due to dizziness. The test has a total possible score of 100 points, whereby 16-34 = mild handicap, 36-52 = moderate handicap, and 54+ = severe handicap.

SECONDARY OUTCOMES:
Balance Error Scoring System (BESS) | At baseline (before the first intervention session) and post-intervention (following the final intervention session)
  The BESS is an objective and quantitative measure used to assess postural stability deficits in mTBI. The assessment will take place on a force plate (BTrackS; balancetrackingsystems.com) in order to measure the participant's center of gravity and sway. The BESS consists of 3 eyes-closed stances: feet together with hands on the hips, single-leg stance on nondominant foot with hands on the hips, and tandem stance with nondominant foot behind the dominant foot. The dominant foot will be identified by determining which foot is used to kick a ball. Each stance is performed on a stable surface (hard floor) and an unstable surface (foam pad) with the eyes closed for 20-seconds per trial. Errors are counted during each trial. BESS results will be reported as a score from 0 to 60, with higher scores representing greater deficits in postural stability (worse outcome).
Activities-Specific Balance Confidence (ABC) Scale | At baseline (before the first intervention session) and post-intervention (following the final intervention session)
  This questionnaire will be used to evaluate participants' balance confidence. An average of balance confidence as it relates to 16 specific everyday activities will be reported from 0% (no confidence) to 100% (complete confidence).
Rivermead Post Concussion Symptoms Questionnaire (RPSQ-3 and RPSQ-13) | At baseline (before the first intervention session) and post-intervention (following the final intervention session)
  This questionnaire will assess the presence and severity of a wide range of post-concussion symptoms.
PROMIS-29 | At baseline (before the first intervention session) and post-intervention (following the final intervention session)
  This questionnaire will assess six domains of health (physical function, anxiety, depression, fatigue, sleep disturbance, social activities) as they relate to participants' dizziness. Questions under the headings "Pain Intensity" and "Pain Interference" will be omitted from this questionnaire as they do not relate to the population.
Motor evoked potential (MEP) | At baseline (before the first intervention session) and post-intervention (following the final intervention session)
  This measure will be used to assess changes in corticospinal excitability. To obtain MEP, thirty individual pulses of TMS at 120% RMT will be applied over the motor hotspot of the dominant hand FDI muscle.
Cytokines (IL-1ß, IL-6, TNF-⍺, IL-10) | At baseline (before the first intervention session) and post-intervention (following the final intervention session)
  A blood sample will be used to evaluate changes in serum concentrations (pg/mL) of cytokines IL-1ß, IL-6, TNF-⍺, IL-10.
C-reactive protein | At baseline (before the first intervention session) and post-intervention (following the final intervention session)
  A blood sample will be used to evaluate changes in serum C-reactive protein concentrations (µg/mL).
Monocyte chemoattractant protein-1 | At baseline (before the first intervention session) and post-intervention (following the final intervention session)
  A blood sample will be used to evaluate changes in serum concentrations (pg/mL) of monocyte chemoattractant protein-1.
Brain-derived neurotrophic factor | At baseline (before the first intervention session) and post-intervention (following the final intervention session)
  A blood sample will be used to evaluate changes in serum concentrations (ng/mL) of brain-derived neurotrophic factor.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Greenbank Concussion Clinic, Hamilton, Ontario
  - McMaster University, Hamilton, Ontario

REFERENCES:
- [Background] Zhao X, Li Y, Tian Q, Zhu B, Zhao Z. Repetitive transcranial magnetic stimulation increases serum brain-derived neurotrophic factor and decreases interleukin-1beta and tumor necrosis factor-alpha in elderly patients with refractory depression. J Int Med Res. 2019 May;47(5):1848-1855. doi: 10.1177/0300060518817417. Epub 2019 Jan 7. PMID 30616482
- [Background] Zuo C, Cao H, Feng F, Li G, Huang Y, Zhu L, Gu Z, Yang Y, Chen J, Jiang Y, Wang F. Repetitive transcranial magnetic stimulation exerts anti-inflammatory effects via modulating glial activation in mice with chronic unpredictable mild stress-induced depression. Int Immunopharmacol. 2022 Aug;109:108788. doi: 10.1016/j.intimp.2022.108788. Epub 2022 Apr 30. PMID 35504201
- [Background] Velioglu HA, Hanoglu L, Bayraktaroglu Z, Toprak G, Guler EM, Bektay MY, Mutlu-Burnaz O, Yulug B. Left lateral parietal rTMS improves cognition and modulates resting brain connectivity in patients with Alzheimer's disease: Possible role of BDNF and oxidative stress. Neurobiol Learn Mem. 2021 Apr;180:107410. doi: 10.1016/j.nlm.2021.107410. Epub 2021 Feb 18. PMID 33610772
- [Background] Rajkumar RP. Immune-inflammatory markers of response to repetitive transcranial magnetic stimulation in depression: A scoping review. Asian J Psychiatr. 2024 Jan;91:103852. doi: 10.1016/j.ajp.2023.103852. Epub 2023 Nov 29. PMID 38070319
- [Background] Cha B, Kim J, Kim JM, Choi JW, Choi J, Kim K, Cha J, Kim M. Therapeutic Effect of Repetitive Transcranial Magnetic Stimulation for Post-stroke Vascular Cognitive Impairment: A Prospective Pilot Study. Front Neurol. 2022 Mar 22;13:813597. doi: 10.3389/fneur.2022.813597. eCollection 2022. PMID 35392634
- [Background] Visser K, Koggel M, Blaauw J, van der Horn HJ, Jacobs B, van der Naalt J. Blood-based biomarkers of inflammation in mild traumatic brain injury: A systematic review. Neurosci Biobehav Rev. 2022 Jan;132:154-168. doi: 10.1016/j.neubiorev.2021.11.036. Epub 2021 Nov 23. PMID 34826510
- [Background] Liao LY, Zhu Y, Peng QY, Gao Q, Liu L, Wang QH, Gao SH, Tao Y, Huang H, Xu PD, Gao CY. Intermittent Theta-Burst Stimulation for Stroke: Primary Motor Cortex Versus Cerebellar Stimulation: A Randomized Sham-Controlled Trial. Stroke. 2024 Jan;55(1):156-165. doi: 10.1161/STROKEAHA.123.044892. Epub 2023 Nov 30. PMID 38037225
- [Background] Paxman E, Stilling J, Mercier L, Debert CT. Repetitive transcranial magnetic stimulation (rTMS) as a treatment for chronic dizziness following mild traumatic brain injury. BMJ Case Rep. 2018 Nov 5;2018:bcr2018226698. doi: 10.1136/bcr-2018-226698. PMID 30396889
- [Background] Zhang JJ, Bai Z, Fong KNK. Priming Intermittent Theta Burst Stimulation for Hemiparetic Upper Limb After Stroke: A Randomized Controlled Trial. Stroke. 2022 Jul;53(7):2171-2181. doi: 10.1161/STROKEAHA.121.037870. Epub 2022 Mar 23. PMID 35317611
- [Background] Platz T, Adler-Wiebe M, Roschka S, Lotze M. Enhancement of motor learning by focal intermittent theta burst stimulation (iTBS) of either the primary motor (M1) or somatosensory area (S1) in healthy human subjects. Restor Neurol Neurosci. 2018;36(1):117-130. doi: 10.3233/RNN-170774. PMID 29439364
- [Background] Huang YZ, Sommer M, Thickbroom G, Hamada M, Pascual-Leonne A, Paulus W, Classen J, Peterchev AV, Zangen A, Ugawa Y. Consensus: New methodologies for brain stimulation. Brain Stimul. 2009 Jan;2(1):2-13. doi: 10.1016/j.brs.2008.09.007. Epub 2008 Oct 7. PMID 20633398
- [Background] Szturm T, Betker AL, Moussavi Z, Desai A, Goodman V. Effects of an interactive computer game exercise regimen on balance impairment in frail community-dwelling older adults: a randomized controlled trial. Phys Ther. 2011 Oct;91(10):1449-62. doi: 10.2522/ptj.20090205. Epub 2011 Jul 28. PMID 21799138
- [Background] Rosiak O, Krajewski K, Woszczak M, Jozefowicz-Korczynska M. Evaluation of the effectiveness of a Virtual Reality-based exercise program for Unilateral Peripheral Vestibular Deficit. J Vestib Res. 2018;28(5-6):409-415. doi: 10.3233/VES-180647. PMID 30714985
- [Background] Smolka W, Smolka K, Markowski J, Pilch J, Piotrowska-Seweryn A, Zwierzchowska A. The efficacy of vestibular rehabilitation in patients with chronic unilateral vestibular dysfunction. Int J Occup Med Environ Health. 2020 Apr 30;33(3):273-282. doi: 10.13075/ijomeh.1896.01330. Epub 2020 Mar 26. PMID 32235946
- [Background] Aligene K, Lin E. Vestibular and balance treatment of the concussed athlete. NeuroRehabilitation. 2013;32(3):543-53. doi: 10.3233/NRE-130876. PMID 23648608
- [Background] Murray DA, Meldrum D, Lennon O. Can vestibular rehabilitation exercises help patients with concussion? A systematic review of efficacy, prescription and progression patterns. Br J Sports Med. 2017 Mar;51(5):442-451. doi: 10.1136/bjsports-2016-096081. Epub 2016 Sep 21. PMID 27655831
- [Background] Broglio SP, Collins MW, Williams RM, Mucha A, Kontos AP. Current and emerging rehabilitation for concussion: a review of the evidence. Clin Sports Med. 2015 Apr;34(2):213-31. doi: 10.1016/j.csm.2014.12.005. Epub 2015 Jan 24. PMID 25818710
- [Background] Toglia JU, Rosenberg PE, Ronis ML. Posttraumatic dizziness; vestibular, audiologic, and medicolegal aspects. Arch Otolaryngol. 1970 Nov;92(5):485-92. doi: 10.1001/archotol.1970.04310050067010. No abstract available. PMID 5506059
- [Background] Hall CD, Herdman SJ, Whitney SL, Anson ER, Carender WJ, Hoppes CW, Cass SP, Christy JB, Cohen HS, Fife TD, Furman JM, Shepard NT, Clendaniel RA, Dishman JD, Goebel JA, Meldrum D, Ryan C, Wallace RL, Woodward NJ. Vestibular Rehabilitation for Peripheral Vestibular Hypofunction: An Updated Clinical Practice Guideline From the Academy of Neurologic Physical Therapy of the American Physical Therapy Association. J Neurol Phys Ther. 2022 Apr 1;46(2):118-177. doi: 10.1097/NPT.0000000000000382. PMID 34864777
- [Background] Ciorba A, Bianchini C, Scanelli G, Pala M, Zurlo A, Aimoni C. The impact of dizziness on quality-of-life in the elderly. Eur Arch Otorhinolaryngol. 2017 Mar;274(3):1245-1250. doi: 10.1007/s00405-016-4222-z. Epub 2016 Jul 22. PMID 27450383
- [Background] Marshall S, Bayley M, McCullagh S, Velikonja D, Berrigan L, Ouchterlony D, Weegar K; mTBI Expert Consensus Group. Updated clinical practice guidelines for concussion/mild traumatic brain injury and persistent symptoms. Brain Inj. 2015;29(6):688-700. doi: 10.3109/02699052.2015.1004755. Epub 2015 Apr 14. PMID 25871303
- [Background] Dougherty JM, Carney M, Hohman MH, Emmady PD. Vestibular Dysfunction. 2023 Jul 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK558926/ PMID 32644352
- [Background] Hartvigsen J, Boyle E, Cassidy JD, Carroll LJ. Mild traumatic brain injury after motor vehicle collisions: what are the symptoms and who treats them? A population-based 1-year inception cohort study. Arch Phys Med Rehabil. 2014 Mar;95(3 Suppl):S286-94. doi: 10.1016/j.apmr.2013.07.029. PMID 24581914
- [Background] Corwin DJ, Wiebe DJ, Zonfrillo MR, Grady MF, Robinson RL, Goodman AM, Master CL. Vestibular Deficits following Youth Concussion. J Pediatr. 2015 May;166(5):1221-5. doi: 10.1016/j.jpeds.2015.01.039. Epub 2015 Mar 5. PMID 25748568
- [Background] Gianoli GJ. Post-concussive Dizziness: A Review and Clinical Approach to the Patient. Front Neurol. 2022 Jan 4;12:718318. doi: 10.3389/fneur.2021.718318. eCollection 2021. PMID 35058868
- [Background] Ryan LM, Warden DL. Post concussion syndrome. Int Rev Psychiatry. 2003 Nov;15(4):310-6. doi: 10.1080/09540260310001606692. PMID 15276952
- [Background] Cassidy JD, Carroll LJ, Peloso PM, Borg J, von Holst H, Holm L, Kraus J, Coronado VG; WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. Incidence, risk factors and prevention of mild traumatic brain injury: results of the WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. J Rehabil Med. 2004 Feb;(43 Suppl):28-60. doi: 10.1080/16501960410023732. PMID 15083870
- [Background] Duprat R, Desmyter S, Rudi de R, van Heeringen K, Van den Abbeele D, Tandt H, Bakic J, Pourtois G, Dedoncker J, Vervaet M, Van Autreve S, Lemmens GM, Baeken C. Accelerated intermittent theta burst stimulation treatment in medication-resistant major depression: A fast road to remission? J Affect Disord. 2016 Aug;200:6-14. doi: 10.1016/j.jad.2016.04.015. Epub 2016 Apr 19. PMID 27107779
- [Background] Hays RD, Spritzer KL, Schalet BD, Cella D. PROMIS(R)-29 v2.0 profile physical and mental health summary scores. Qual Life Res. 2018 Jul;27(7):1885-1891. doi: 10.1007/s11136-018-1842-3. Epub 2018 Mar 22. PMID 29569016
- [Background] King NS, Crawford S, Wenden FJ, Moss NE, Wade DT. The Rivermead Post Concussion Symptoms Questionnaire: a measure of symptoms commonly experienced after head injury and its reliability. J Neurol. 1995 Sep;242(9):587-92. doi: 10.1007/BF00868811. PMID 8551320
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Bell DR, Guskiewicz KM, Clark MA, Padua DA. Systematic review of the balance error scoring system. Sports Health. 2011 May;3(3):287-95. doi: 10.1177/1941738111403122. PMID 23016020
- [Background] Jacobson GP, Newman CW. The development of the Dizziness Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1990 Apr;116(4):424-7. doi: 10.1001/archotol.1990.01870040046011. PMID 2317323